CLINICAL TRIAL: NCT06862349
Title: The Effect of Propofol Induction Using Total Body Weight and Lean Body Weight Obtained by Tomographic Measurements; on the Depth of Anesthesia in Patients Receiving General Anesthesia
Brief Title: Propofol Induction Based on Lean Body Weight on the Depth of Anesthesia
Acronym: propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: propofol induction
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Propofol Adverse Reaction
Keywords: lean body mass; propofol adverse reaction; general anaesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): All patients were taken to the operating room, and in addition to routine monitoring, BIS and SedLine monitoring were provided. All patients received 1 mcg/kg of fentanyl. Group T received propofol at a dose of 2-2.5 mg/kg based on total body weight. The laryngeal mask will be placed once an adequate depth of anesthesia is achieved.
  Interventions: Drug: Group T received propofol at a dose of 2-2.5 mg/kg based on total body weight
- Group L (Active Comparator): All patients were taken to the operating room, and in addition to routine monitoring, BIS and SedLine monitoring were provided. All patients received 1 mcg/kg of fentanyl. Group T received propofol at a dose of 2-2.5 mg/kg based on lean body weight. The laryngeal mask will be placed once an adequate depth of anesthesia is achieved.
  Interventions: Drug: Group L received propofol at 2-2,5mg/kg dose based on lean body weight, which was calculated from CT imaging by a radiologist.

INTERVENTIONS:
Drug: Group T received propofol at a dose of 2-2.5 mg/kg based on total body weight — A total of 120 patients undergoing general anesthesia for urological surgeries at our hospital were included in the study. Patients were randomized into two groups (Group T/Group L). All patients were taken to the operating room, and in addition to routine monitoring, BIS and SedLine monitoring were provided. All patients received 1 mcg/kg of fentanyl. Group T received propofol at a dose of 2-2.5 mg/kg based on total body weight. Propofol was administered at a rate of 100 mg/min. The laryngeal mask will be placed once an adequate depth of anesthesia is achieved. All data were recorded at 2-minute intervals for 6 minutes before and after induction. The collected data were statistically analyzed for comparison.
  Arms: Group T
Drug: Group L received propofol at 2-2,5mg/kg dose based on lean body weight, which was calculated from CT imaging by a radiologist. — A total of 120 patients undergoing general anesthesia for urological surgeries at our hospital were included in the study. Patients were randomized into two groups (Group T/Group L). All patients were taken to the operating room, and in addition to routine monitoring, BIS and SedLine monitoring were provided. All patients received 1 mcg/kg of fentanyl. Group L received propofol at 2-2,5mg/kg dose based on lean body weight, which was calculated from CT imaging by a radiologist. Propofol was administered at a rate of 100 mg/min. The laryngeal mask will be placed once an adequate depth of anesthesia is achieved. All data were recorded at 2-minute intervals for 6 minutes before and after induction. The collected data were statistically analyzed for comparison.
  Arms: Group L

SUMMARY:
Propofol has significant hemodynamic side effects. It is a lipophilic agent and is generally used at a dose of 2-2.5 mg/kg for induction. In patients with a body mass index (BMI) greater than 25, it can lead to serious complications. This patient group often has comorbidities such as hypertension, coronary artery disease, left ventricular hypertrophy, stroke, and obstructive sleep apnea.

Hemodynamic profile changes are influenced by both the rate of propofol administration and the total dose. Therefore, it is necessary to investigate the appropriate dose and infusion rate of propofol during anesthesia induction.

The primary aim of this study is to compare the effects of propofol induction doses, determined based on total body weight and lean body weight (calculated using tomography), on anesthesia depth using BIS and SedLine monitoring in patients with BMI >25.

The secondary aim of the study is to compare propofol induction doses calculated using two different methods in terms of:

* Mean arterial pressure (MAP),
* Frequency of hypotension (MAP <65),
* Frequency of Trendelenburg position or vasopressor requirement and their response,
* Tachycardia (heart rate >100 bpm),
* Frequency of hypertension (SBP >140).

Additionally, the sensitivity and delay rates of BIS and SedLine monitoring in determining anesthesia depth were compared.

A total of 120 patients undergoing general anesthesia for urological surgeries at our hospital were included in the study. Patients were randomized into two groups (Group T/Group L). All patients were taken to the operating room, and in addition to routine monitoring, BIS and SedLine monitoring were provided. All patients received 1 mcg/kg of fentanyl.

* Group T received propofol at a dose of 2-2.5 mg/kg based on total body weight.
* Group L received propofol at a dose of 2-2.5 mg/kg based on lean body weight, which was calculated from CT imaging by a radiologist.
* Propofol was administered at a rate of 100 mg/min.

The laryngeal mask will be placed once an adequate depth of anesthesia is achieved.

All data were recorded at 2-minute intervals for 6 minutes before and after induction. The collected data were statistically analyzed for comparison.

ELIGIBILITY:
Inclusion Criteria:

* A total of 120 patients of both genders,
* Aged 18-65 years,
* BMI >25
* Scheduled for elective surgery under general anesthesia in the urology operating room

Exclusion Criteria:

* Patients under 18 years of age or over 65 years old
* Patients unable to read, understand, or sign the consent form
* Hemodynamically unstable patients
* Patients with contraindications to anesthetic drugs
* Patients who do not wish to participate in the study
* Patients deemed unsuitable by the researcher
* Patients with advanced dementia or behavioral disorders
* Patients using psychiatric medications or abusing drugs
* Patients requiring awake intubation
* Emergency surgical procedures
* Patients with more than a 5% weight change between the time of the CT scan --and the surgery day
* A time gap of more than 2 months between the CT scan and the surgery day

The criteria for discontinuing the study are as follows:

* Patients who develop anaphylaxis
* Airway failure
* Patients who develop unexpected complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
anaesthesia debt | 30 minute
  Anesthesia depth was assessed using BIS and SedLine monitoring before and after induction and recorded every 2 minutes.

SECONDARY OUTCOMES:
mean arterial pressure | 30 minute
  Mean arterial pressure was measured before and after induction and recorded every 2 minutes.
trendelenburg | 30 minute
  The need for Trendelenburg position due to hypotension before and after induction was recorded every 2 minutes.
vasopressor | 30 minute
  The need for vasopressor due to hypotension before and after induction was recorded every 2 minutes.
heart | 30 minute
  Heart rate was recorded every 2 minutes before and after induction, allowing the rate of tachycardia development to be monitored as a study outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmidt GN, Bischoff P, Standl T, Lankenau G, Hilbert M, Schulte Am Esch J. Comparative evaluation of Narcotrend, Bispectral Index, and classical electroencephalographic variables during induction, maintenance, and emergence of a propofol/remifentanil anesthesia. Anesth Analg. 2004 May;98(5):1346-53, table of contents. doi: 10.1213/01.ane.0000111209.44119.30. PMID 15105213
- [Result] Gurses E, Sungurtekin H, Tomatir E, Dogan H. Assessing propofol induction of anesthesia dose using bispectral index analysis. Anesth Analg. 2004 Jan;98(1):128-131. doi: 10.1213/01.ANE.0000090314.43496.1D. PMID 14693603
- [Result] Pilge S, Zanner R, Schneider G, Blum J, Kreuzer M, Kochs EF. Time delay of index calculation: analysis of cerebral state, bispectral, and narcotrend indices. Anesthesiology. 2006 Mar;104(3):488-94. doi: 10.1097/00000542-200603000-00016. PMID 16508396
- [Result] Rusch D, Arndt C, Eberhart L, Tappert S, Nageldick D, Wulf H. Bispectral index to guide induction of anesthesia: a randomized controlled study. BMC Anesthesiol. 2018 Jun 15;18(1):66. doi: 10.1186/s12871-018-0522-8. PMID 29902969